CLINICAL TRIAL: NCT02267005
Title: The Effect of Creatine Supplementation on Muscle Function in Childhood Myositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Brian Feldman, Division Head, Rheumatology / Sr Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 1000041466
Record Dates: First submitted 2014-10-01; First posted 2014-10-17 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Juvenile Dermatomyositis
MeSH Terms: conditions — Dermatomyositis | interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): patients on this arm will be treated with creapure supplements
  Interventions: Dietary Supplement: Creapure
- Placebo (Placebo Comparator): patients on this arm will be given a placebo glucose tablet supplement
  Interventions: Dietary Supplement: Glucose Tablet

INTERVENTIONS:
Dietary Supplement: Creapure — Patients will be prescribed a creapure supplement by weight, to be taken 3x/day for the duration of the trial. They will be randomized to an active product start time using a multiple baseline design.
  Other Names: ultrapure creatine monohydrate
  Arms: Treatment
Dietary Supplement: Glucose Tablet — Patients will be prescribed the placebo supplement by weight, to be taken 3x/day for the duration of the trial. They will be randomized to an active product start time using a multiple baseline design.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This project will bring together a multidisciplinary team of pediatric rheumatologists, neurologists, metabolic geneticists and exercise physiologists to determine the effect of creatine (CR) supplementation on muscle function and muscle metabolism in children with Dermatomyositis (DM). The investigators propose using well-established exercise testing techniques as well as new, powerful exercise imaging protocols in order to better delineate the effects of CR on muscle pathophysiology in a non-invasive way. Evidence from this study will provide information regarding the effect of creatine supplementation on muscle function in DM. Improvements in muscle function and fatigue through CR use may also contribute to an improvement in quality of life and have significant clinical implications for the treatment of children with DM.

ELIGIBILITY:
Inclusion Criteria:

* Ages 7 to 18 years
* Diagnosis of probable JDM (onset <16 years) according to Bohan and Peter criteria
* Subjects on a stable course of medication (unlikely to change over study treatment period as determined by the treating physician)
* Minimum height of 132.5cm

Exclusion Criteria:

* Subjects newly diagnosed with JDM within the previous 6 months
* Subjects unable to cooperate with study procedures, or too weak to participate in the exercise testing
* Subjects with impaired kidney function as determined from baseline visit screening lab values
* Subjects who are currently pregnant or planning to become pregnant within the study period
* Subjects who are shorter than 132.5cm

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2015-03; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Muscle function | 6 months
  Will be determined by mean power output using a Wingate cycle ergometer protocol

SECONDARY OUTCOMES:
Muscle metabolism | 6 months
  The effects of creatine supplementation on key metabolites responsible for proper energy shuttling in healthy muscle will be measured at rest and using exercise protocols in subjects with P-MRS.
Quality of life | 6 months
  Both overall and health-related quality of life will be measured at each study visit with the Quality of My Life scale.
Disease Activity | 6 months
  Will be measured using the International Myositis Assessment and Clinical Studies Group (IMACS) before and after creatine supplementation
Muscle Strength | 6 months
  Will be estimated at each study visit from a maximal jump test and hand grip strength.
Fatigue | 6 months
  Will be determined using the PedsQL fatigue module which has been validated for use in children with fibromyalgia and rheumatic disease.
Adherence | 6 months
  This will be assessed based on a positive blood plasma and urine tests for creatine use over the course of the study period, amount of medication remaining and through self-reports using study diaries.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada